CLINICAL TRIAL: NCT02397330
Title: the Association of Ultrasound Guided Suprascapular and Supraclavicular Nerve Block Provides Adequate Analgesia in Comparison With Ultrasound Guided Interscalene Block
Brief Title: is There an Alternative to Ultrasound Guided Interscalene Block?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tunisian Military Hospital (Other)
Responsible Party: Principal Investigator, Dr trabelsi walid, associate professor, MD, Tunisian Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TunisianMH1
Record Dates: First submitted 2015-03-09; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Regional Anesthesia; Interscalene Block; Shoulder Surgery
MeSH Terms: interventions — Bupivacaine; Ultrasonography; Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- group BIS (Active Comparator): scheduled for ultrasound guided interscalene blockade with 30 ml of bupivacaine 0.25%
  Interventions: Drug: bupivacaine; Device: ultrasound; Drug: morphine
- group BS (Experimental): scheduled for selective blockade of the ultrasound guided suprascapular (15 ml bupivacaine 0.25%) and supraclavicular (15 ml bupivacaine 0.25%) nerves blocks
  Interventions: Drug: bupivacaine; Device: ultrasound; Drug: morphine

INTERVENTIONS:
Drug: bupivacaine
Device: ultrasound — ultrasound guided nerve blocks
Drug: morphine

SUMMARY:
Interscalene brachial plexus block is the gold standard for perioperative pain management in shoulder surgery. However, this technique would have side effects and potential serious complications. The aim of this study is to compare between the combination of ultrasound guided suprascapular and supraclavicular nerve blocks versus ultrasound guided interscalene brachial plexus block for post operative analgesia after shoulder instability surgery with latarjet procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* 18-75 years of age, inclusive
* shoulder surgery (LATARJET technique)

Exclusion Criteria:

* contraindications to brachial plexus block (e.g., allergy to local anesthetics, coagulopathy, malignancy or infection in the area)
* existing neurological deficit
* pregnancy
* history of neck surgery or radiotherapy
* severe respiratory disease
* inability to understand the informed consent and demands of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Visual Analogic Scale | until 48 hours postoperative
  quality of postoperative analgesia

SECONDARY OUTCOMES:
time to perform the blocks | up to 5 minutes
patient satisfaction | 48 hours post performing nerves blocks
  scale from 0 (not satisfied at all) to 100 (full satisfaction)
occurrence of complications | 48 hours post performing nerves blocks
total dose of morphine consumption in mg | during 48 hours post operative

REFERENCES:
- [Derived] Trabelsi W, Ben Gabsia A, Lebbi A, Sammoud W, Labbene I, Ferjani M. Suprascapular block associated with supraclavicular block: An alternative to isolated interscalene block for analgesia in shoulder instability surgery? Orthop Traumatol Surg Res. 2017 Feb;103(1):77-83. doi: 10.1016/j.otsr.2016.10.012. Epub 2016 Dec 2. PMID 27916737